CLINICAL TRIAL: NCT03969303
Title: Comparison Between Retinal Images Captured by NOTAL-OCT V2.5 and Zeiss Cirrus / Heidelberg Spectralis SD OCT - Study Protocol
Brief Title: NOTAL-OCT V.2.5 vs Commercial OCT in AMD Patients
Status: Completed | Type: Observational
Sponsor: Notal Vision Ltd. (Industry)
Collaborators: Elman Retina Group (Other)
Responsible Party: Sponsor
Organization: Notal Vision Inc. (Industry)
Other Study IDs: C2018.008
Record Dates: First submitted 2018-10-23; First posted 2019-05-31 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-10

CONDITIONS: AMD - Age-Related Macular Degeneration; Diabetic Macular Edema
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NOTAL OCT v.2.5 and Commercial OCT on AMD Patients: OCT Images will be obtained in the central 10 degrees of the macula in AMD patients using the NOTAL OCT v.2.5 device and a Commercial device (Zeiss Cirrus/Heidelberg SPECTRALIS).
  Interventions: Device: Notal Vision Optical Coherence Tomography Device Version 2.5 (NOTAL-OCT V2.5)

INTERVENTIONS:
Device: Notal Vision Optical Coherence Tomography Device Version 2.5 (NOTAL-OCT V2.5) — OCT SCAN

SUMMARY:
Primary objective:

To evaluate the level of agreement between the NOTAL-OCT V2.5 and a commercial OCT in the presence of fluid as identified in the OCT images, in the central 10 degrees of the macula in AMD (Age-related Macular Degeneration) patients.

Secondary objectives:

1. To evaluate the level of agreement between the NOTAL-OCT V2.5 and a commercial OCT in the presence of fluid as identified in the OCT images, in the central 10 degrees of the macula in DME (Diabetic Macular Edema) patients.
2. To evaluate patient experience when self-operating the Notal-OCT V2.5.

DETAILED DESCRIPTION:
To evaluate the sensitivity and specificity regarding the presence and absence of fluid on OCT images of AMD patients. OCT images from the central 10 degrees of the macula in AMD patients will be obtained using the NOTAL OCT v.2.5 and a commercial OCT device (Zeiss Cirrus / Heidlberg SPECTRALIS). These images will be evaluated for the presence/absence of fluid in the images by a human grader. The sensitivity and specificity will be determined by comparison of the presence/absence of fluid in the NOTAL OCT v2.5 images with the presence/absence of fluid in the commercial OCT images.

To evaluate the sensitivity and specificity regarding the presence and absence of fluid on OCT images of DME patients. OCT images from the central 10 degrees of the macula in DME patients will be obtained using the NOTAL OCT v.2.5 and a commercial OCT device (Zeiss Cirrus / Heidlberg SPECTRALIS). These images will be evaluated for the presence/absence of fluid in the images by a human grader. The sensitivity and specificity will be determined by comparison of the presence/absence of fluid in the NOTAL OCT v2.5 images with the presence/absence of fluid in the commercial OCT images.

Patients will complete a questionnaire regarding the usability of the NOTAL-OCT v.2.5 device

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to give informed consent (IC)
* 18 years of age or older
* Diagnosis of AMD (age-related macular degeneration) and/or DME (diabetic macular edema) in the study eye as confirmed by the investigator and recorded in the patient's clinical record
* Ability to undergo OCT (optical coherence tomography) testing
* Visual acuity of 20/400 Snellen (6/120) or better in the study eye

Exclusion Criteria:

- Any ophthalmic or systemic condition that in the opinion of the investigator would preclude the patient from participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AMD and DME patients
Sampling Method: Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2018-10-20 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-10-04 (Actual)

PRIMARY OUTCOMES:
Comparison of presence/absence of fluid on OCT images from NOTAL-OCT v.2.5 device with a commercial OCT device, in AMD (Age-related Macular Degeneration) patients | less than an hour
  To evaluate the sensitivity and specificity regarding the presence and absence of fluid on OCT images of AMD patients. OCT images from the central 10 degrees of the macula in AMD patients will be obtained using the NOTAL OCT v.2.5 and a commercial OCT device (Zeiss Cirrus / Heidlberg SPECTRALIS). These images will be evaluated for the presence/absence of fluid in the images by a human grader. The sensitivity and specificity will be determined by comparison of the presence/absence of fluid in the NOTAL OCT v2.5 images with the presence/absence of fluid in the commercial OCT images.

SECONDARY OUTCOMES:
Comparison of presence/absence of fluid on OCT images from NOTAL-OCT v.2.5 device with a commercial OCT device, in DR (Diabetic Retinopathy) patients | less then an hour
  To evaluate the sensitivity and specificity regarding the presence and absence of fluid on OCT images of DR patients. OCT images from the central 10 degrees of the macula in DR patients will be obtained using the NOTAL OCT v.2.5 and a commercial OCT device (Zeiss Cirrus / Heidlberg SPECTRALIS). These images will be evaluated for the presence/absence of fluid in the images by a human grader. The sensitivity and specificity will be determined by comparison of the presence/absence of fluid in the NOTAL OCT v2.5 images with the presence/absence of fluid in the commercial OCT images.
Patient experience using the NOTAL-OCT v.2.5 device | less than an hour
  Patients will complete a questionnaire with 13 statements or questions regarding the usability of the NOTAL-OCT v.2.5 device. For the first 10 statements, patients are asked to specify a level of agreement to the statement. The scale is named "Level of Agreement" and ranges from 1 = strongly agree, to 5 = strongly disagree. A patient's indicating a value of 1 is considered to be a better outcome. The remaining 3 questions are free-form.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Elman, Principal Investigator — Michael Elman, M.D. 9114 Philadelphia Rd #310 Baltimore, Maryland 21237
Locations (1):
- Elman Retina Group, PA, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided